INFORMED VOLUNTARY CONSENT FORM

Dear participant,

This survey aims to collect information about the effect of EMDR on pain in Rheumatoid Arthritis patients within the scope of the research titled "Effect of eye movement desensitization and reprocessing (EMDR) on pain in rheumatoid arthritis patients". The results will help determine the

effect of EMDR on pain.

There are 14 questions in the survey. Your response time to the questions is on average 5 minutes. Participation in the research is on a voluntary basis. If you wish, you can leave the research at any time during the research, provided that you inform the principal researcher. Any records that reveal your identity will be kept confidential and will not be made public. Only people other than you who have direct access to your medical records (such as the Ethics Committee that approves the research, other than those on the research team) will know that you have participated in this study. However, as at every stage of the study, all your information will be kept confidential even when the results of the study are published. The accuracy of your answers to the questions in the questionnaire is very important in terms of the quality of the research. Therefore, we ask you to answer the questions in the

survey correctly, and thank you for your cooperation.

Specialist Nurse Müjde MORAN

**Health Sciences Institute** 

Mental Health and Diseases Nursing

Department Ph.D. Student

Tel: 05055774978

PERSONAL INFORMATION FORM

"Effect of eye movement desensitization and reprocessing (EMDR) on pain in rheumatoid arthritis patients"

| Date:/ |
|---------------------------------------------|
| Patient's Name and Surname: |
| Phone number: |
| Working group: ( ) Control ( ) Intervention |
| 1. Your age: |
| 2. Your gender: ( ) Female ( ) Male |

3. Your marital status: ( ) Married ( ) Single

| 4. Your education status: |
|---|
| ( )Not literate ( )Literate ( )Primary/secondary school graduate ( )High school graduate |
| ( )University graduate ()Graduate |
| 5. What is your income status according to you? |
| ( ) Income less than expenses |
| ( ) Income equal to expenses |
| ( ) Income more than expenses |
| 6. Do you know about EMDR? ( ) Yes ( ) No |
| 7. If your answer to the sixth question is yes, where did you get this information? |
| 8. Has EMDR been applied before? ( ) Yes No |
| 9. How long ago were you diagnosed with Rheumatoid Arthritis? monthyear |
| 10. Do you have a chronic disease other than this one? ( ) Yes (please specify) ( ) No |
| 11. How often do you have pain per week? |
| ( ) None |
| ( ) Very little |
| ( ) 1-2 times a week |
| ( ) Often |
| 12. How long does it usually last when you have pain?minuteshoursdays |
| 13. Do you use regular painkillers when you have pain? ( ) Yes ( ) No |
| 14. Which of the options is more suitable for your ability to perform your daily living activities? |
| ( ) I can do it independently |
| ( ) Painful but able to perform |
| ( ) I am at a level to continue some activities |
| ( ) I am addicted |